CLINICAL TRIAL: NCT06120361
Title: The Swedish BioFINDER - Primary Care Study
Acronym: ADetect
Status: Recruiting | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Erik Stomrud, M.D., PhD, Skane University Hospital
Other Study IDs: ADetect
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Mild Dementia; Mild Cognitive Impairment; SCD; Alzheimer Disease; Lewy Body Disease; Frontotemporal Degeneration; Vascular Dementia
Keywords: Primary care, early diagnosis, blood, biomarkers, cognitive testing
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Lewy Body Disease; Dementia, Vascular; Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients in primary care with cognitive symptoms
  Interventions: Diagnostic Test: Plasma APS 2 score; Diagnostic Test: Plasma p-tau217/np-tau217; Diagnostic Test: Plasma p-tau217; Diagnostic Test: Plasma neurofilament light (NfL); Diagnostic Test: Plasma Ab42/Ab40; Diagnostic Test: MRI and CT of the brain; Diagnostic Test: Different cognitive tests

INTERVENTIONS:
Diagnostic Test: Plasma APS 2 score — APS 2 score (combination of ptau217/nptau217 and Ab42/Ab40). The cut off will be predefined. The samples will be analysed prospectively every two weeks.
Diagnostic Test: Plasma p-tau217/np-tau217 — The cut off will be predefined. The samples will be analysed prospectively every two weeks.
Diagnostic Test: Plasma p-tau217 — The cut off will be predefined. The samples will be analysed prospectively every two weeks.
Diagnostic Test: Plasma neurofilament light (NfL) — The cut off will be predefined. The samples will be analysed prospectively every two weeks.
Diagnostic Test: Plasma Ab42/Ab40 — The cut off will be predefined. The samples will be analysed prospectively every two weeks.
Diagnostic Test: MRI and CT of the brain — Structural brain imaging
Diagnostic Test: Different cognitive tests — Both standard paper-and-pen tests as well as digital cognitive tests will be evaluated.

SUMMARY:
The overall aim of the study is to improve the diagnostic accuracy of AD and cognitive impairment in primary care settings to ensure better care and treatment as well as facilitate correct referrals to specialized memory clinics. The investigators will strive to recruit diverse and representative populations of patients with subjective cognitive decline (SCD), mild cognitive impairment (MCI) and mild dementia. The specific aims of the study are to:

1. Improve the detection of mild cognitive impairment (MCI) and dementia in primary care.
2. Develop and evaluate cognitive tests, blood-based biomarkers and brain imaging methods that are suitable for accurate and early diagnosis of Alzheimer's disease (AD) in primary care.
3. To prospectively validate plasma AD biomarkers for diagnosis of patients with cognitive symptoms who are evaluated in primary care.
4. Determine whether blood AD biomarkers improve patient management in primary care.

DETAILED DESCRIPTION:
AIMS

The overall aim of the study is to improve the diagnostic accuracy of AD and cognitive impairment in primary care settings to ensure better care and treatment as well as facilitate correct referrals to specialized memory clinics. The investigators will strive to recruit diverse and representative populations of patients with subjective cognitive decline (SCD), mild cognitive impairment (MCI) and mild dementia. The specific aims of the study are to:

1. Improve the detection of mild cognitive impairment (MCI) and dementia in primary care.

   Early detection of cognitive impairment can lead to improved care, optimized treatments, and highlight issues regarding decision making, incorrect utilizations of healthcare resources and driving ability.Despite this, primary care still uses the same tools as 30-40 years ago, which have a low sensitivity for MCI. In this project, the investigators will identify the optimal cognitive screening tests by doing head-to-head comparisons of novel and traditional cognitive tests including computerized tests and smartphone apps that can run daily tests of memory and executive function.
2. Develop and evaluate cognitive tests, blood-based biomarkers and brain imaging methods that are suitable for accurate and early diagnosis of Alzheimer's disease (AD) in primary care.

   AD is the most common dementia (causing about 70% of all dementia cases) and there are currently 4 registered symptomatic treatments that improve cognition, activities of daily function and may delay the time to nursing homes. Detection of AD is therefore essential in order to start the treatment. Further, promising trials suggest that disease-modifying AD treatments might be available in the future targeting Aβ (the cause and hallmark pathology of AD). In this scenario, it essential that AD is identified at an early stage before neurodegeneration is wide-spread. To tackle this, the investigators will develop and validate methods that can accurately detect people with early AD in a primary care setting, including i) cognitive screening tests (e.g. computerized tests and smartphone apps); ii) novel blood-based biomarkers (e.g. mass spectrometry based plasma p-tau217 and Ab42/40 measures as well as the combination of these two biomarkers in C2N Diagnostics' PrecivityAD2 test), and iii) widely available brain imaging methods (including a comparison between computed tomography scan [CT] and Magnetic resonance imaging scan [MRI]). The ultimate goal is to develop brief and cost-effective diagnostic algorithms. The investigators will both validate a previous algorithm that the investigators have published as well as test new ones, including the PrecivityAD2 test result known as the Amyloid Probability Score 2 (APS2, ranging from 0-100 for the likelihood of brain amyloid plaques).
3. To prospectively validate plasma AD biomarkers for diagnosis of patients with cognitive symptoms who are evaluated in primary care. The investigators here intend to study the clinical robustness and accuracy of plasma AD biomarkers in real-world settings by using high-performing plasma assays over a 2-3 year time period. In this study, plasma samples are collected as part of clinical praxis and analyzed on a bi-weekly basis throughout the study period (and not in single batches). The investigators will (1) use pre-defined cut offs for each biomarker (similar to real world clinical practice), and (2) use an accurate reference standard (i.e., cerebrospinal fluid (CSF)/Positron emission tomography (PET) AD biomarkers). The effects of potential confounders (such as kidney function) on diagnostic accuracy will also be studied. The investigators will only use really top-performing plasma assays for each biomarker including for p-tau217 and Ab42/Ab40.
4. Determine whether blood AD biomarkers improve patient management in primary care.

   As often noted by regulatory authorities, it is important to know if novel diagnostic methods improve the actual management of patients in real world settings. Consequently, the investigators study whether the most promising plasma biomarkers for symptomatic AD (including the APS2) will improve AD diagnosis beyond what is currently done as part of clinical practice. The physician will document the most likely diagnosis (and the certainty of the diagnosis) after having performed an interview with the patient and informant, as well as evaluated the patient's cognitive test results, routine blood tests and structural brain imaging. The physician will then re-evaluate the diagnosis (and certainty of diagnosis) after having obtained the APS2, plasma p-tau217 and Ab42/Ab40 results, and the pre- and post-test diagnosis will be compared to the reference standard (i.e. presence of AD brain pathology as determined with biomarkers). Change in treatment and care of the patient after evaluating blood-based biomarkers will also be recorded similar to how amyloid-PET was evaluated in the IDEAS study.

   PARTICIPANTS

   The study will consecutively recruit 1200 patients seeking medical care due to mild cognitive symptoms in primary care units. They will be recruited at approximately 20-30 primary care facilities in Skåne. The patients will as usual first meet a general practitioner who performs a basic investigation of the patient to rule out other obvious causes causing the cognitive symptoms other than a dementia disorder, such as depression, sleep deprivation, etc. The patients, whose cognitive symptoms are not clearly explained by psychiatric or somatic conditions, will be assessed with cognitive tests by a dementia nurse or occupational therapist at the primary care unit.

   ASSESSMENTS AT THE PRIMARY CARE UNIT

   At the primary care units, the investigators will collect data to be able to design optimal and cost-effective diagnostic algorithms for dementia disorder, especially AD. In order to do that the investigators will perform different cognitive tests, including smartphone-based tests, to determine impairment of global cognition as well as different cognitive domains. Informed consent is signed before the study begins.

   i) Cognitive Testing at the primary care unit The primary care tests are summarized below. These include tradition and novel pen and paper tests, iPad tests, smartphone-based tests for home-based testing and the use of a digital pen.

   The Montreal Cognitive Assessment (MoCA)

   Mini-Mental State Examination (MMSE)

   The 10-word list from the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) (immediate, delayed and recognition recall)

   Symbol Digit Modalities Test (SDMT)

   Animal Fluency

   Cube copying

   The clock drawing test

   Immediate and delayed recall of pictures test

   Trail Making Test A and B

   Mini-Cog

   CANTAB Paired Associate Learning (iPad)

   CANTAB Reaction Time (iPad)

   Mezurio Gallery game (smartphone)

   Mezurio Tilt Task (smartphone)

   Digital Clock Test

   Speech recognition tests (ki elements)

   In-house developed iPad test battery

   Cognitive Function Instrument (CFI)

   Amsterdam iADL scale

   ii) Blood sampling at the primary care unit Recent breakthroughs by our group and others show that it is possible to accurately detect cerebral Aβ and tau using blood-based biomarkers. Blood will be collected in 10 mL EDTA tubes, which are centrifuged (2000g) within 1 hour. Plasma will then be aliquoted into LoBind tubes and sent by ordinary transport to the Clinical Chemistry unit either in Malmö or Lund for storage at -80°C. Some of these plasma samples will be analysed prospectively every two weeks.

   iii) Brain imaging ordered by the primary care unit A short a short MRI examination and a CT scan of the brain will be ordered by the primary care unit, and performed at the local hospital. The brain atrophy pattern may reveal the type of underlying dementia disorder that is the cause of cognitive symptoms.

   iv) Assessment of change in management and diagnosis After the initial basic dementia investigation (current clinical practice) the primary care physician will 1) note the most likely diagnosis of the patient, 2) rate his/her confidence in the diagnosis of the patient and 3) note the plans for further investigations and treatment. Thereafter, the clinician will get access to the newly developed APS2 diagnostic algorithm that includes prospectively measured plasma p-tau217 ratio and Ab42/40 levels). After obtaining the results of the APS2 algorithm the medical doctor will again 1) note the most likely diagnosis of the patient, 2) rate his/her confidence in the diagnosis of the patient and 3) note the plans for further investigations and treatment. This will allow us to evaluate what impact the new cognitive and blood tests have on physicians' decision making and if the clinical diagnostic accuracy was improved.

   ESTABLISHMENT OF THE STANDARD OF TRUTH - ASSESSMENT OF THE MEMORY CLINIC

   After the visit at the primary care unit, the patient will be referred to the Memory Clinic to determine the cognitive function and clinical diagnosis, which will be blinded to all investigations done at the primary care unit (besides the CT scan). The following will be performed:
   1. Extensive cognitive testing by an experienced neuropsychologist using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) neuropsychological battery that does not overlap with the cognitive tests at the primary care units. These tests are done according to clinical routine practice at our Memory clinic.
   2. Cognitive, neurological and psychiatric assessments by a physician specialized in cognitive disorders. These assessments are done according to clinical routine practice at our Memory clinic.
   3. Detection of brain amyloid pathology by either cerebrospinal fluid AD biomarkers (CSF Aβ42/Aβ40 [Lumipulse; Fujirebio] and CSF p-tau217 [Eli Lilly]), alternatively 18F-flutemetamol PET will be used if there are contraindications for lumbar puncture. These assessments are done according to clinical routine practice at our Memory clinic.

   A consensus diagnosis will be established based on the neuropsychological, medical history, and CSF data (blinded to the cognitive test data from the primary care unit and the blood-based biomarker data). Analysis of CSF Aβ42/Aβ40 [Lumipulse; Fujirebio] and CSF p-tau217 [Eli Lilly] will be used to determine if the patient is AD pathology negative or positive (alternatively amyloid PET if there are contraindications for LP).

   Patients will also be followed over 3-5 years to determine the rate of cognitive decline and progression to AD dementia in those with either SCD or MCI at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. The patient seeks medical help because of cognitive symptoms experienced by the patient and/or informant OR The general practitioner suspects a progressive neurodegenerative disorder including, but not limited to, Alzheimer's disease, Lewy body disease, frontotemporal lobar degeneration or subcortical vascular cognitive impairment.
2. The main symptom is usually memory complaints, but could also be executive, visuo-spatial, language, or attention complaints.
3. Age ≥40 years
4. Subjective cognitive decline, mild cognitive impairment or mild dementia

Exclusion Criteria:

1. Already diagnosed dementia
2. Significant unstable systemic illness or organ failure that makes it difficult to participate.
3. Current significant alcohol or substance misuse.
4. Refusing investigation at the Memory clinic
5. Cognitive impairment with acute onset due to stroke
6. The cognitive impairment can with certainty be explained by another condition or disease such as significant anemia, infection, severe sleep deprivation, psychotic disorder, moderate-severe depression, alcohol abuse etc.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will consecutively recruit 1200 patients seeking medical care due to mild cognitive symptoms in primary care units. They will be recruited at approximately 20-30 primary care facilities in Skåne. The patients will as usual first meet a general practitioner who performs a basic investigation of the patient to rule out other obvious causes causing the cognitive symptoms other than a dementia disorder, such as depression, sleep deprivation, etc. The patients, whose cognitive symptoms are not clearly explained by psychiatric or somatic conditions, will be assessed with cognitive tests by a dementia nurse or occupational therapist at the primary care unit.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of brain AD pathology as determined by CSF AD biomarkers | At baseline (cross-sectional)
  CSF Ab42/Ab40 and p-tau217

SECONDARY OUTCOMES:
Clinical diagnosis supported by CSF biomarkers | At baseline (cross-sectional)
  Clinical diagnosis based on The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) but supported by CSF biomarkers
Presence of brain AD pathology as determined by amyloid PET imaging | At baseline (cross-sectional)
  Amyloid PET imaging
Presence of brain AD pathology as determined by tau PET imaging | At baseline (cross-sectional)
  Tau PET imaging
Rate of progression to AD dementia in patients with SCD or MCI at baseline | Follow-up over appr. 4 years
  Development of AD dementia during follow-up diagnosed using DSM-5 and supported by CSF biomarkers
Change in patient management | At baseline (cross-sectional)
  Change in suggested diagnosis, treatment, referral or ordered diagnostic tests
Change in diagnostic confidence | At baseline (cross-sectional)
  Change in diagnostic confidence of the treating physician

CONTACTS AND LOCATIONS:
Locations (1):
- Primary care centers in Region Skåne, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within one year after study completion